CLINICAL TRIAL: NCT06611137
Title: SBRT Followed by Chemoimmunotherapy of Toripalimab Plus Docetaxel and Cisplatin for Larynx Preservation in Patients with Locally Regionally Advanced Squamous Cell Carcinoma of the Larynx and Hypopharynx
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-373-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Laryngeal Cancer; Hypopharynx Cancer
Keywords: SBRT; immunotherapy; larynx preservation; laryngeal cancer; hypopharynx cancer
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT+Toripalimab Plus Docetaxel and Cisplatin (Experimental): SBRT for gross tumor and metastatic lymph nodes, followed by neoadjuvant chemoimmunotherapy of Toripalimab Plus Docetaxel and Cisplatin
  Interventions: Combination Product: SBRT+Toripalimab Plus Docetaxel and Cisplatin

INTERVENTIONS:
Combination Product: SBRT+Toripalimab Plus Docetaxel and Cisplatin — All participants will receive SBRT (18Gy/3 fractions, QOD ) to gross tumor and metastatic lymph nodes, followed by neoadjuvant chemoimmunotherapy of Toripalimab (240mg) Plus Docetaxel (75mg/m2, q3w) and Cisplatin (75mg/m2, q3w) for 3 cycles. If tumor has complete or partial response at 2 weeks after the last course of neoadjuvant chemotherapy, participants will then receive intensity modulated radiotherapy (54Gy/27 fractions). If tumor is stable or progressive, participants will receive radical resection with or without postoperative intensity modulated radiotherapy when necessary.

SUMMARY:
This trial aims to evaluate the safety and efficiency of SBRT followed by Chemoimmunotherapy of Toripalimab Plus Docetaxel and Cisplatin for Patients with Locally Regionally Advanced Squamous Cell Carcinoma of the Larynx and Hypopharynx

ELIGIBILITY:
Inclusion Criteria:

* Laryngeal (T3-4N0-3M0 ) and hypopharyngeal ( T2-4N0-3M0) cancers staged by AJCC8th
* age 18-70
* PS score 0-1
* normal functions to tolerate chemotherapy, immunotherapy and radiotherapy

Exclusion Criteria:

* Patients with a combination of other malignant tumours
* Individuals with contraindications to immunotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
objective response rate | two weeks after the last course of neoadjuvant chemotherapy
  complete and partial response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided